CLINICAL TRIAL: NCT01644643
Title: An Open-Label, Randomized, Multicenter, Phase III Study of Ceftazidime Avibactam (CAZ-AVI, Formerly CAZ104) and Best Available Therapy for the Treatment of Infections Due to Ceftazidime Resistant Gram Negative Pathogens
Brief Title: Ceftazidime-Avibactam for the Treatment of Infections Due to Ceftazidime Resistant Pathogens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4280C00006; 2012-000726-21
Record Dates: First submitted 2012-06-28; First posted 2012-07-19 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Complicated Urinary Tract Infection; Complicated Intra-abdominal Infection
Keywords: Ceftazidime,; avibactam,; metronidazone,; Anti-Infectives
MeSH Terms: interventions — avibactam, ceftazidime drug combination; Metronidazole

ARMS (2):
- Ceftazidime - Avibactam ( CAZ-AVI) (Experimental): IV treatment
  Interventions: Drug: Ceftazidime - Avibactam ( CAZ-AVI); Drug: Metronidazole
- Best Available Therapy (Active Comparator): IV treatment
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: Ceftazidime - Avibactam ( CAZ-AVI) — Ceftazidime 2000 mg and 500 mg of avibactam Patients randomized to receive CAZ-AVI will receive an infusion of CAZ-AVI (2000 mg ceftazidime and 500 mg avibactam) every 8 hours administered by intravenous (IV) infusion in a volume of 100 mL at a constant rate over 120 minutes
  Arms: Ceftazidime - Avibactam ( CAZ-AVI)
Drug: Best Available Therapy — Patients randomized to receive Best Available Therapy will receive the best available standard of care (SOC) anti-infective therapy for their infection administered in accord with approved local label recommendation
  Arms: Best Available Therapy
Drug: Metronidazole — Anti-infective, 500 mg (cIAI only) Patients randomized to receive CAZ-AVI for cIAI will also receive metronidazole (500 mg) administered by IV infusion in a volume of 100 mL at a constant rate over 60 minutes immediately following the CAZ-AVI infusion
  Other Names: Flagyl
  Arms: Ceftazidime - Avibactam ( CAZ-AVI)

SUMMARY:
To Evaluate the Effects of Ceftazidime-Avibactam and Best Available Therapy in patients with complicated urinary tract infections and complicated intra-abdominal infections.

DETAILED DESCRIPTION:
An Open-Label, Randomized, Multicenter, Phase III Study of Ceftazidime Avibactam (CAZ-AVI, formerly CAZ104) and Best Available Therapy for the Treatment of Infections Due to Ceftazidime Resistant Gram Negative Pathogens

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥18 and ≤90 years of age
* Female patients can participate if they are surgically sterile or completed menopause or females capable of having children and agree not to attempt pregnancy while receiving IV study therapy and for a period of 7 days after
* Patient has a ceftazidime-resistant Gram negative pathogen that was isolated from an appropriate culture within 5 days prior to study entry (ie, within 5 days prior to Screening; the study-qualifying culture), which was determined to be the causative agent of the entry infection

Exclusion Criteria:

* Patient has an APACHE II score >30 (cIAI patients only)
* Patient has an infection due to Gram negative pathogen that is unlikely to respond to CAZ-AVI treatment (eg, Acinetobacter spp., Stenotrophomonas spp.)
* Patient is receiving hemodialysis or peritoneal dialysis or had a renal transplant Patient is immunocompromised
* Patient has a rapidly progressive or terminal illness with a high risk of mortality due to any cause, including acute hepatic failure, respiratory failure or severe septic shock such that they are unlikely to survive the 4- to 5-week study period.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newell, MBBS, MRCP, Study Director — AstraZeneca
Locations (43):
- United States (2):
  - Research Site, Shreveport, Louisiana
  - Research Site, Lima, Ohio
- Argentina (2):
  - Research Site, El Talar
  - Research Site, La Plata
- Bulgaria (6):
  - Research Site, Pazardzhik
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
- Croatia (2):
  - Research Site, Slavonski Brod
  - Research Site, Zagreb
- Research Site, Prague, Czechia
- Research Site, Tours, France
- Israel (4):
  - Research Site, Nazareth
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Mexico (2):
  - Research Site, Guadalajara
  - Research Site, Mexico City
- Peru (2):
  - Research Site, Cusco
  - Research Site, Surco
- Research Site, Manila, Philippines
- Research Site, Szczecin, Poland
- Research Site, Bucharest, Romania
- Russia (6):
  - Research Site, Irkutsk
  - Research Site, Krasnodar
  - Research Site, Novosibirsk
  - Research Site, Penza
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Research Site, Johannesburg, South Africa
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Diyarbakır
  - Research Site, Istanbul
- Ukraine (4):
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Zaporizhzhya

REFERENCES:
- [Background] Carmeli Y, Armstrong J, Laud PJ, Newell P, Stone G, Wardman A, Gasink LB. Ceftazidime-avibactam or best available therapy in patients with ceftazidime-resistant Enterobacteriaceae and Pseudomonas aeruginosa complicated urinary tract infections or complicated intra-abdominal infections (REPRISE): a randomised, pathogen-directed, phase 3 study. Lancet Infect Dis. 2016 Jun;16(6):661-673. doi: 10.1016/S1473-3099(16)30004-4. Epub 2016 Apr 20. PMID 27107460
- [Derived] Torres A, Wible M, Tawadrous M, Irani P, Stone GG, Quintana A, Debabov D, Burroughs M, Bradford PA, Kollef M. Efficacy and safety of ceftazidime/avibactam in patients with infections caused by beta-lactamase-producing Gram-negative pathogens: a pooled analysis from the Phase 3 clinical trial programme. J Antimicrob Chemother. 2023 Nov 6;78(11):2672-2682. doi: 10.1093/jac/dkad280. PMID 37700689
- [Derived] Cheng K, Newell P, Chow JW, Broadhurst H, Wilson D, Yates K, Wardman A. Safety Profile of Ceftazidime-Avibactam: Pooled Data from the Adult Phase II and Phase III Clinical Trial Programme. Drug Saf. 2020 Aug;43(8):751-766. doi: 10.1007/s40264-020-00934-3. PMID 32602065
- [Derived] Mendes RE, Castanheira M, Woosley LN, Stone GG, Bradford PA, Flamm RK. Characterization of beta-Lactamase Content of Ceftazidime-Resistant Pathogens Recovered during the Pathogen-Directed Phase 3 REPRISE Trial for Ceftazidime-Avibactam: Correlation of Efficacy against beta-Lactamase Producers. Antimicrob Agents Chemother. 2019 May 24;63(6):e02655-18. doi: 10.1128/AAC.02655-18. Print 2019 Jun. PMID 30910899
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- [Derived] Nichols WW, Stone GG, Newell P, Broadhurst H, Wardman A, MacPherson M, Yates K, Riccobene T, Critchley IA, Das S. Ceftazidime-Avibactam Susceptibility Breakpoints against Enterobacteriaceae and Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e02590-17. doi: 10.1128/AAC.02590-17. Print 2018 Nov. PMID 30061279
- [Derived] Stone GG, Newell P, Gasink LB, Broadhurst H, Wardman A, Yates K, Chen Z, Song J, Chow JW. Clinical activity of ceftazidime/avibactam against MDR Enterobacteriaceae and Pseudomonas aeruginosa: pooled data from the ceftazidime/avibactam Phase III clinical trial programme. J Antimicrob Chemother. 2018 Sep 1;73(9):2519-2523. doi: 10.1093/jac/dky204. PMID 29912399
- [Derived] Stone GG, Bradford PA, Newell P, Wardman A. In Vitro Activity of Ceftazidime-Avibactam against Isolates in a Phase 3 Open-Label Clinical Trial for Complicated Intra-Abdominal and Urinary Tract Infections Caused by Ceftazidime-Nonsusceptible Gram-Negative Pathogens. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e01820-16. doi: 10.1128/AAC.01820-16. Print 2017 Feb. PMID 27872067
- Available data/document: Study Protocol: D4280C00006 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1452&filename=Clinical%20Study%20Protocol_3%20Redacted%20amended.pdf — D4280C00006 Clinical Study Protocol
- Available data/document: Study Protocol: D4280C00006 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1452&filename=Clinical%20Study%20Protocol%20Amendment%202%20Redacted%20amended.pdf — D4280C00006 Clinical Study Protocol Amendment 2 Redacted amended
- Available data/document: Study Protocol: D4280C00006 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1452&filename=Clinical%20Study%20Protocol%20Amendment%203%20Redacted%20amended.pdf — D4280C00006 Clinical Study Protocol Amendment 3 Redacted amended

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 333 patients were randomized in 53 centers in 16 countries: 306 patients had complicated urinary tract infection (cUTI) and 27 patients had complicated intra-abdominal infection (cIAI). The first patient was randomized on 07JAN2013 and the last patient was randomized on 29AUG2014. One patient in CAZ-AVI arm didn't receive study drug.
Groups:
- cIAI:Best Available Therapy: cIAI: Best Available Therapy Determinated by Investigator
- cIAI:CAZ-AVI + Metronidazole: cIAI:CAZ-AVI (2000 mg ceftazidime/500 mg avibactam) plus metronidazole (500 mg)
- cUTI:Best Available Therapy: cUTI:Best Available Therapy Determinated by Investigator
- cUTI:CAZ-AVI: cUTI: CAZ-AVI
Period: Overall Study
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Started | 15 | 12 | 153 | 153
Completed | 13 | 12 | 148 | 143
Not Completed | 2 | 0 | 5 | 10
Not completed — Death | 1 | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1
Not completed — Other Eligibility criteria | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Microbiological modified intent to treat: all patients who have a diagnosis of cIAI or cUTI with a ceftazidime-resistant Gram-negative pathogen on the study-qualifying culture and who received at least 1 dose of study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI | Total
Number analyzed (Participants) | 11 | 10 | 137 | 144 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (11.12) [50 to 86] | 49.9 (16.14) [26 to 73] | 61.3 (15.33) [18 to 90] | 64.3 (14.64) [18 to 88] | 62.6 (15.12) [18 to 90]
Age, Customized [Number; unit: Participants]
  18-45 Years | 0 | 3 | 21 | 19 | 43
  46-64 Years | 3 | 5 | 49 | 41 | 98
  65-74 Years | 4 | 2 | 40 | 46 | 92
  75-90 Years | 4 | 0 | 27 | 38 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 63 | 64 | 137
  Male | 7 | 4 | 74 | 80 | 165
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 0 | 1 | 2 | 3
  Black Or African American | 0 | 1 | 1 | 2 | 4
  Other | 0 | 0 | 4 | 4 | 8
  White | 11 | 9 | 131 | 136 | 287

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at Test of Cure (TOC) in Microbiological Modified Intent-to-treat (mMITT) Analysis Set
Description: Proportion of patients with clinical cure at the TOC visit in the mMITT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Groups:
- cUTI:CAZ-AVI: cUTI:CAZ-AVI (2000 mg ceftazidime/500 mg avibactam)
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Clinical cure | 6 [27.0 to 80.0] | 8 [86.3 to 95.4] | 129 [89.3 to 97.2] | 132
  Clinical failure | 0 | 0 | 2 | 2
  Indeterminate | 5 | 2 | 6 | 10

2. Secondary Outcome: Clinical Response at End of Treatment (EOT) in mMITT Analysis Set.
Description: Proportion of patients with clinical cure at the EOT visit in the mMITT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 28 hours after completion of last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Clinical cure | 6 | 9 | 136 | 142
  Clinical failure | 0 | 0 | 0 | 0
  Indeterminate | 5 | 1 | 1 | 2

3. Secondary Outcome: Clinical Response at Follow-up 1 (FU1) in mMITT Analysis Set
Description: Proportion of patients with clinical cure at the FU1 visit in the mMITT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: cIAI: 27-37 calendar days from randomization/cUTI: 20-27 calendar days from randomization
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Clinical cure | 6 | 8 | 121 | 127
  Clinical failure | 0 | 0 | 8 | 5
  Indeterminate | 5 | 2 | 8 | 12

4. Secondary Outcome: Clinical Response at Follow-up 2 (FU2) in mMITT Analysis Set
Description: Proportion of patients with clinical cure at the FU2 visit in the mMITT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: At FU2, data was only collected for the cUTI Arms: 28-34 calendar days from randomization
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 0 | 0 | 137 | 144
Participant
  Clinical cure |  |  | 118 | 123
  Clinical failure |  |  | 13 | 11
  Indeterminate |  |  | 6 | 10

5. Secondary Outcome: Clinical Response at EOT in Extended Microbiologically Evaluable (EME) at EOT Analysis Set.
Description: Proportion of patients with clinical cure at the EOT visit in the EME at EOT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 28 hours after completion of last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Extended Microbiological Evaluable at EOT analysis set.
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 9 | 127 | 134
Participant
  Clinical cure | 5 | 9 | 127 | 134
  Clinical failure | 0 | 0 | 0 | 0

6. Secondary Outcome: Clinical Response at TOC in EME at TOC Analysis Set.
Description: Proportion of patients with clinical cure at the TOC visit in the EME at TOC analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 6-12 days after last infusion of study therapy.Duration of study therapy was 5 to 21 days.
Population: Extended Microbiological Evaluable at TOC analysis set.
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 8 | 122 | 128
Participant
  Clinical cure | 5 | 8 | 120 | 126
  Clinical failure | 0 | 0 | 2 | 2

7. Secondary Outcome: Clinical Response at FU1 in EME at FU1 Analysis Set.
Description: Proportion of patients with clinical cure at the FU1 visit in EME at FU1 analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: cIAI: 27-37 calendar days from randomization/cUTI: 20-27 calendar days from randomization
Population: Extended Microbiological Evaluable at FU1 analysis set.
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 7 | 118 | 124
Participant
  Clinical cure | 5 | 7 | 110 | 120
  Clinical failure | 0 | 0 | 8 | 4

8. Secondary Outcome: Clinical Response at FU2 in EME at FU2 Analysis Set
Description: Proportion of patients with clinical cure at the FU2 visit in EME at FU2 analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary.
Time Frame: At FU2, data was only collected for the cUTI Arms: 28-34 calendar days from randomization
Population: Extended Microbiological Evaluable at FU2 analysis set.
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 0 | 0 | 114 | 116
Participant
  Clinical cure |  |  | 102 | 106
  Clinical failure |  |  | 12 | 10

9. Secondary Outcome: Clinical Cure at TOC by Baseline Gram-negative Pathogen in mMITT Analysis Set
Description: Proportion of patients with clinical cure at TOC visit by baseline pathogen (>=10% of frequency in the combined cIAI and cUTI patients) in the mMITT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 6-12 days after last infusion of study therapy.Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  E. coli - Clinical cure (n=6, 4, 57, 59) | 2 | 3 | 54 | 53
  K. pneumoniae - Clinical cure (n=3, 5, 65, 55) | 2 | 3 | 61 | 54
  P. aeruginosa - clinical cure (n=1, 1, 5, 14) | 1 | 1 | 5 | 12

10. Secondary Outcome: Clinical Cure at TOC by Baseline Gram-negative Pathogen in EME at TOC Analysis Set
Description: Proportion of patients with clinical cure at TOC visit by baseline Gram-negative pathogen (>=10% of frequency in the combined cIAI and cUTI patients) in EME at TOC analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 6-12 days after last infusion of study therapy.Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at TOC
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 8 | 124 | 131
Participant
  E. coli - Clinical cure (n=2, 3, 48, 52) | 2 | 3 | 47 | 51
  K. pneumoniae - Clinical cure (n=2, 3, 59, 53) | 2 | 3 | 59 | 53
  P. aeruginosa - Clinical cure (n=1, 1, 5, 12) | 1 | 1 | 5 | 12

11. Secondary Outcome: Clinical Cure at TOC by Previously Failed Treatment Class in mMITT Analysis Set
Description: Proportion of patients with clinical cure at TOC visit by previously failed treatment class in the mMITT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  At least 1 failed - Clin. cure (n=4,7,12,7) | 3 | 7 | 12 | 6
  Antibiotics - Clin. cure (n=0,1,0,0) | 0 | 1 | 0 | 0
  Carbapenems - Clin. cure (n=1,0,1,2) | 0 | 0 | 1 | 1
  Comb of Sulf/Trime inc Deriv-Clin. cure(n=0,0,2,0) | 0 | 0 | 2 | 0
  Combs Of Peni. Inc B-Lact. Inhib.-Cure(n=1,3,0,2) | 1 | 3 | 0 | 2
  Cortico,Po. Comb W/Antibio.-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  First-Gen. Cephalosporins-Clin. cure (n=0,0,2,0) | 0 | 0 | 2 | 0
  Fluoroquinolones - Clin. cure (n=1,2,7,1) | 0 | 2 | 7 | 1
  Glycopeptide Antibacterials-Clin. cure (n=1,0,0,0) | 0 | 0 | 0 | 0
  Imidazole Derivatives - Clin. cure (n=2,3,0,0) | 1 | 3 | 0 | 0
  Other Aminoglycosides-Clin. cure (n=0,0,1,1) | 0 | 0 | 1 | 1
  Other Antibacterials-Clin. cure (n=0,1,1,0) | 0 | 1 | 1 | 0
  Other Antibio. F. Topic. Use-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  Penici. With Ext. Spectrum-Clin. cure(n=0,1,0,0) | 0 | 1 | 0 | 0
  Third-Gen.Cephalosporins -Clin. cure(n=2,4,3,2) | 2 | 4 | 3 | 2

12. Secondary Outcome: Clinical Cure at EOT by Previously Failed Treatment Class in EME at EOT Analysis Set
Description: Proportion of patients with clinical cure at EOT visit by previously failed treatment class in EME at EOT analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 28 hours after completion of last infusion of study therapy.Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at EOT
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 9 | 127 | 134
Participant
  Antibiotics - Clin. cure (n=0,1,0,0) | 0 | 1 | 0 | 0
  Carbapenems - Clin. cure (n=0,0,1,1) | 0 | 0 | 1 | 1
  Comb of Sulf/Trime inc Deriv-Clin. cure(n=0,0,2,0) | 0 | 0 | 2 | 0
  Combs Of Peni. Inc B-Lact. Inhib.-Cure(n=1,3,0,2) | 1 | 3 | 0 | 2
  Cortico,Po. Comb W/Antibio.-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  First-Gen. Cephalosporins-Clin. cure (n=0,0,2,0) | 0 | 0 | 2 | 0
  Fluoroquinolones - Clin. cure (n=0,2,5,1) | 0 | 2 | 5 | 1
  Imidazole Derivatives - Clin. cure (n=1,3,0,0) | 1 | 3 | 0 | 0
  Other Aminoglycosides-Clin. cure (n=0,0,1,1) | 0 | 0 | 1 | 1
  Other Antibacterials-Clin. cure (n=0,1,1,0) | 0 | 1 | 1 | 0
  Other Antibio. F. Topic. Use-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  Penici. With Ext. Spectrum-Clin. cure(n=0,1,0,0) | 0 | 1 | 0 | 0
  Third-Gen.Cephalosporins -Clin. cure(n=2,4,2,2) | 2 | 4 | 2 | 2

13. Secondary Outcome: Clinical Cure at TOC by Previously Failed Treatment Class in EME at TOC Analysis Set
Description: Proportion of patients with clinical cure at TOC visit by previously failed treatment class in EME at TOC analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at TOC
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 8 | 122 | 128
Participant
  Antibiotics - Clin. cure (n=0,1,0,0) | 0 | 1 | 0 | 0
  Carbapenems - Clin. cure (n=0,0,1,1) | 0 | 0 | 1 | 1
  Comb of Sulf/Trime inc Deriv-Clin. cure(n=0,0,2,0) | 0 | 0 | 2 | 0
  Combs Of Peni. Inc B-Lact. Inhib.-Cure(n=1,3,0,2) | 1 | 3 | 0 | 2
  Cortico,Po. Comb W/Antibio.-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  First-Gen. Cephalosporins-Clin. cure (n=0,0,2,0) | 0 | 0 | 2 | 0
  Fluoroquinolones - Clin. cure (n=0,2,5,1) | 0 | 2 | 5 | 1
  Imidazole Derivatives - Clin. cure (n=1,3,0,0) | 1 | 3 | 0 | 0
  Other Aminoglycosides-Clin. cure (n=0,0,0,1) | 0 | 0 | 0 | 1
  Other Antibacterials-Clin. cure (n=0,1,1,0) | 0 | 1 | 1 | 0
  Other Antibio. F. Topic. Use-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  Penici. With Ext. Spectrum-Clin. cure(n=0,1,0,0) | 0 | 1 | 0 | 0
  Third-Gen.Cephalosporins -Clin. cure(n=2,4,2,2) | 2 | 4 | 2 | 2

14. Secondary Outcome: Clinical Cure at FU1 by Previously Failed Treatment Class in EME at FU1 Analysis Set
Description: Proportion of patients with clinical cure at FU1 visit by previously failed treatment class in EME at FU1 analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary; for cIAI patients no drainage or surgical intervention after 96 hours from randomization is necessary (ie. drainage or surgical intervention up to 96 hours from randomization is permissible).
Time Frame: cIAI: 27-37 calendar days from randomization/cUTI: 20-27 calendar days from randomization
Population: Extended microbiologically evaluable at FU1
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 7 | 118 | 124
Participant
  Antibiotics - Clin. cure (n=0,1,0,0) | 0 | 1 | 0 | 0
  Carbapenems - Clin. cure (n=0,0,1,1) | 0 | 0 | 1 | 1
  Comb of Sulf/Trime inc Deriv-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  Combs Of Peni. Inc B-Lact. Inhib.-Cure(n=1,3,0,2) | 1 | 3 | 0 | 2
  Cortico,Po. Comb W/Antibio.-Clin. cure(n=0,0,1,0) | 0 | 0 | 0 | 0
  First-Gen. Cephalosporins-Clin. cure (n=0,0,2,0) | 0 | 0 | 2 | 0
  Fluoroquinolones - Clin. cure (n=0,2,5,1) | 0 | 2 | 4 | 1
  Imidazole Derivatives - Clin. cure (n=1,3,0,0) | 1 | 3 | 0 | 0
  Other Aminoglycosides-Clin. cure (n=0,0,0,1) | 0 | 0 | 0 | 1
  Other Antibacterials-Clin. cure (n=0,1,1,0) | 0 | 1 | 1 | 0
  Other Antibio. F. Topic. Use-Clin. cure(n=0,0,1,0) | 0 | 0 | 1 | 0
  Penici. With Ext. Spectrum-Clin. cure(n=0,1,0,0) | 0 | 1 | 0 | 0
  Third-Gen.Cephalosporins -Clin. cure(n=2,4,1,2) | 2 | 4 | 0 | 2

15. Secondary Outcome: Clinical Cure at FU2 by Previously Failed Treatment Class in EME at FU2 Analysis Set
Description: Proportion of patients with clinical cure at FU2 visit by previously failed treatment class in EME at FU2 analysis set. Clinical cure: Complete resolution or significant improvement of signs and symptoms of the index infection such that no further antibacterial therapy (other than those allowed per protocol) is necessary.
Time Frame: At FU2, data was only collected for the cUTI Arms: 28-34 calendar days from randomization
Population: Extended microbiologically evaluable at FU2
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 0 | 0 | 114 | 116
Participant
  Carbapenems - Clin. cure (n=1,0) |  |  | 0 | 0
  Comb of Sulf/Trime inc Deriv-Clin. cure(n=1,0) |  |  | 0 | 0
  Combs Of Peni. Inc B-Lact. Inhib.-Cure(n=0,2) |  |  | 0 | 2
  Cortico,Po. Comb W/Antibio.-Clin. cure(n=1,0) |  |  | 0 | 0
  First-Gen. Cephalosporins-Clin. cure (n=2,0) |  |  | 2 | 0
  Fluoroquinolones - Clin. cure (n=5,0) |  |  | 4 | 0
  Other Aminoglycosides-Clin. cure (n=0,1) |  |  | 0 | 1
  Other Antibacterials-Clin. cure (n=1,0) |  |  | 0 | 0
  Other Antibio. F. Topic. Use-Clin. cure(n=1,0) |  |  | 1 | 0
  Third-Gen.Cephalosporins -Clin. cure(n=1,1) |  |  | 0 | 1

16. Secondary Outcome: Per-patient Microbiological Response at EOT in mMITT Analysis Set
Description: Microbiological responses as per the protocoled criteria: responses other than "indeterminate" were classified as "favorable" or "unfavorable." Favorable microbiological response assessments included "eradication" and "presumed eradication." Unfavorable microbiological response assessments included "persistence," "persistence with increasing minimum inhibitory concentration (MIC)," and "presumed persistence." Indeterminate microbiologic response assessments included cIAI patients where the clinical response was changed to indeterminate due to a Surgical Review Panel assessment of inadequate source control (ie, circumstances that preclude classification as eradication, presumed eradication, persistence, persistence with increasing MIC, and presumed persistence).
Time Frame: 28 hours after completion of last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Favorable | 6 | 9 | 130 | 136
  Unfavorable | 0 | 0 | 1 | 1
  Indeterminate | 5 | 1 | 6 | 7

17. Secondary Outcome: Per-patient Microbiological Response at TOC in mMITT Analysis Set
Description: as for outcome 16
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Favorable | 6 | 8 | 88 | 118
  Unfavorable | 0 | 0 | 42 | 17
  Indeterminate | 5 | 2 | 7 | 9

18. Secondary Outcome: Per-patient Microbiological Response at FU1 in mMITT Analysis Set
Description: as for outcome 16
Time Frame: cUTI: 20-27 calendar days from randomization/cIAI: 27-37 calendar days from randomization
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Favorable | 6 | 8 | 78 | 103
  Unfavorable | 0 | 0 | 50 | 29
  Indeterminate | 5 | 2 | 9 | 12

19. Secondary Outcome: Per-patient Microbiological Response at FU2 in mMITT Analysis Set
Description: as for outcome 16
Time Frame: At FU2, data was only collected for the cUTI Arms: 28-34 calendar days from randomization
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 0 | 0 | 137 | 144
Participant
  Favorable |  |  | 73 | 99
  Unfavorable |  |  | 54 | 35
  Indeterminate |  |  | 10 | 10

20. Secondary Outcome: Per-patient Microbiological Response at EOT in EME at EOT Analysis Set
Description: as for outcome 16
Time Frame: 28 hours after completion of last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at EOT
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 9 | 127 | 134
Participant
  Favorable | 5 | 9 | 127 | 133
  Unfavorable | 0 | 0 | 0 | 1

21. Secondary Outcome: Per-patient Microbiological Response at TOC in EME at TOC Analysis Set
Description: as for outcome 16
Time Frame: 6-12 days after last infusion of study therapy.Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at TOC
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 8 | 124 | 131
Participant
  Favorable | 5 | 8 | 84 | 114
  Unfavorable | 0 | 0 | 40 | 17

22. Secondary Outcome: Per-patient Microbiological Response at FU1 in EME at FU1 Analysis Set
Description: as for outcome 16
Time Frame: cUTI: 20-27 calendar days from randomization/cIAI: 27-37 calendar days from randomization
Population: Extended microbiologically evaluable at FU1
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 7 | 120 | 126
Participant
  Favorable | 5 | 7 | 75 | 98
  Unfavorable | 0 | 0 | 45 | 28

23. Secondary Outcome: Per-patient Microbiological Response at FU2 in EME at FU2 Analysis Set
Description: as for outcome 16
Time Frame: At FU2, data was only collected for the cUTI Arms: 28-34 calendar days from randomization
Population: Extended microbiologically evaluable at FU2
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 0 | 0 | 115 | 117
Participant
  Favorable |  |  | 68 | 85
  Unfavorable |  |  | 47 | 32

24. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at EOT in mMITT Analysis Set
Description: Proportion of patients with a favorable per-pathogen microbiological response for pathogens (>=10% of frequency in the combined cIAI and cUTI patients): favourable microbiological response includes: Eradication Absence (or urine quantification less than 10^4 CFU/ml for cUTI patients) of causative pathogen from an appropriately obtained specimen at the site of infection. If the patient was bacteremic at Screening, the bacteremia has also resolved. Presumed eradication where, repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure (specific to cIAI population).
Time Frame: 28 hours after completion of last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Escherichia coli - Favorable (n=6, 4, 57, 59) | 2 | 3 | 53 | 57
  Escherichia coli - Unfavorable (n=6, 4, 57, 59) | 0 | 0 | 0 | 0
  Escherichia coli - Indeterminate (n=6, 4, 57, 59) | 4 | 1 | 4 | 2
  Kleb. pneumoniae - Favorable (n=3, 5, 65, 55) | 2 | 4 | 61 | 52
  Kleb. pneumoniae - Unfavorable (n=3, 5, 65, 55) | 0 | 0 | 1 | 0
  Kleb. pneumoniae - Indeterminate (n=3, 5, 65, 55) | 1 | 1 | 3 | 3
  Pseudo. aeruginosa - Favorable (n=1, 1, 5, 14) | 1 | 1 | 5 | 14
  Pseudo. aeruginosa - Unfavorable (n=1, 1, 5, 14) | 0 | 0 | 0 | 0
  Pseudo. aeruginosa - Indeterminate (n=1, 1, 5, 14) | 0 | 0 | 0 | 0

25. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at TOC in mMITT Analysis Set
Description: as for outcome 24
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Escherichia coli - Favorable (n=6, 4, 57, 59) | 2 | 3 | 38 | 52
  Escherichia coli - Unfavorable (n=6, 4, 57, 59) | 0 | 0 | 16 | 3
  Escherichia coli - Indeterminate (n=6, 4, 57, 59) | 4 | 1 | 3 | 4
  Kleb. pneumoniae - Favorable (n=3, 5, 65, 55) | 2 | 3 | 43 | 46
  Kleb. pneumoniae - Unfavorable (n=3, 5, 65, 55) | 0 | 0 | 19 | 8
  Kleb. pneumoniae - Indeterminate (n=3, 5, 65, 55) | 1 | 2 | 3 | 1
  Pseudo. aeruginosa - Favorable (n=1, 1, 5, 14) | 1 | 1 | 3 | 11
  Pseudo. aeruginosa - Unfavorable (n=1, 1, 5, 14) | 0 | 0 | 2 | 2
  Pseudo. aeruginosa - Indeterminate (n=1, 1, 5, 14) | 0 | 0 | 0 | 1

26. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at FU1 in mMITT Analysis Set
Description: as for outcome 24
Time Frame: cIAI: 27-37 calendar days from randomization/cUTI: 20-27 calendar days from randomization
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Escherichia coli - Favorable (n=6, 4, 57, 59) | 2 | 3 | 33 | 45
  Escherichia coli - Unfavorable (n=6, 4, 57, 59) | 0 | 0 | 18 | 12
  Escherichia coli - Indeterminate (n=6, 4, 57, 59) | 4 | 1 | 6 | 2
  Kleb. pneumoniae - Favorable (n=3, 5, 65, 55) | 2 | 3 | 39 | 42
  Kleb. pneumoniae - Unfavorable (n=3, 5, 65, 55) | 0 | 0 | 23 | 10
  Kleb. pneumoniae - Indeterminate (n=3, 5, 65, 55) | 1 | 2 | 3 | 3
  Pseudo. aeruginosa - Favorable (n=1, 1, 5, 14) | 1 | 1 | 3 | 8
  Pseudo. aeruginosa - Unfavorable (n=1, 1, 5, 14) | 0 | 0 | 2 | 2
  Pseudo. aeruginosa - Indeterminate (n=1, 1, 5, 14) | 0 | 0 | 0 | 4

27. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at FU2 in mMITT Analysis Set
Description: Proportion of patients with a favorable per-pathogen microbiological response for pathogens (>=10% of frequncy in the combined cIAI and cUTI patients): favourable microbiological response includes: Eradication Absence (or urine quantification less than 10^4 CFU/ml for cUTI patients) of causative pathogen from an appropriately obtained specimen at the site of infection. If the patient was bacteremic at Screening, the bacteremia has also resolved. Presumed eradication where, repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure (specific to cIAI population).
Time Frame: At FU2, data was only collected for the cUTI Arms: 28-34 calendar days from randomization
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 0 | 0 | 137 | 144
Participant
  Escherichia coli - Favorable (n=0, 0, 57, 59) |  |  | 32 | 43
  Escherichia coli - Unfavorable (n=0, 0, 57, 59) |  |  | 19 | 14
  Escherichia coli - Indeterminate (n=0, 0, 57, 59) |  |  | 6 | 2
  Kleb. pneumoniae - Favorable (n=0, 0, 65, 55) |  |  | 35 | 39
  Kleb. pneumoniae - Unfavorable (n=0, 0, 65, 55) |  |  | 26 | 14
  Kleb. pneumoniae - Indeterminate (n=0, 0, 65, 55) |  |  | 4 | 2
  Pseudo. aeruginosa - Favorable (n=0, 0, 5, 14) |  |  | 2 | 10
  Pseudo. aeruginosa - Unfavorable (n=0, 0, 5, 14) |  |  | 3 | 2
  Pseudo. aeruginosa - Indeterminate (n=0, 0, 5, 14) |  |  | 0 | 2

28. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at EOT in EME at EOT Analysis Set
Description: as for outcome 27
Time Frame: 28 hours after completion of last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at EOT
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 9 | 127 | 134
Participant
  Escherichia coli - Favorable (n=2, 3, 51, 55) | 2 | 3 | 51 | 55
  Escherichia coli - Unfavorable (n=2, 3, 51, 55) | 0 | 0 | 0 | 0
  Kleb. pneumoniae - Favorable (n=2, 4, 60, 52) | 2 | 4 | 60 | 52
  Kleb. pneumoniae - Unfavorable (n=2, 4, 60, 52) | 0 | 0 | 0 | 0
  Pseudo. aeruginosa - Favorable (n=1, 1, 5, 14) | 1 | 1 | 5 | 14
  Pseudo. aeruginosa - Unfavorable (n=1, 1, 5, 14) | 0 | 0 | 0 | 0

29. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at TOC in EME at TOC Analysis Set
Description: as for outcome 27
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at TOC
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 8 | 124 | 131
Participant
  Escherichia coli - Favorable (n=2, 3, 49, 53) | 2 | 3 | 34 | 50
  Escherichia coli - Unfavorable (n=2, 3, 49, 53) | 0 | 0 | 15 | 3
  Kleb. pneumoniae - Favorable (n=2, 3, 60, 53) | 2 | 3 | 42 | 45
  Kleb. pneumoniae - Unfavorable (n=2, 3, 60, 53) | 0 | 0 | 18 | 8
  Pseudo. aeruginosa - Favorable (n=1, 1, 5, 13) | 1 | 1 | 3 | 11
  Pseudo. aeruginosa - Unfavorable (n=1, 1, 5, 13) | 0 | 0 | 2 | 2

30. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at FU1 in EME at FU1 Analysis Set
Description: as for outcome 27
Time Frame: cIAI: 27-37 calendar days from randomization/cUTI: 20-27 calendar days from randomization
Population: Extended microbiologically evaluable at FU1
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 7 | 120 | 126
Participant
  Escherichia coli - Favorable (n=2, 3, 46, 54) | 2 | 3 | 30 | 43
  Escherichia coli - Unfavorable (n=2, 3, 46, 54) | 0 | 0 | 16 | 11
  Kleb. pneumoniae - Favorable (n=2, 2, 59, 50) | 2 | 2 | 38 | 40
  Kleb. pneumoniae - Unfavorable (n=2, 2, 59, 50) | 0 | 0 | 21 | 10
  Pseudo. aeruginosa - Favorable (n=1, 1, 5, 10) | 1 | 1 | 3 | 8
  Pseudo. aeruginosa - Unfavorable (n=1, 1, 5, 10) | 0 | 0 | 2 | 2

31. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at FU2 in EME at FU2 Analysis Set
Description: as for outcome 27
Time Frame: At FU2, data was only collected for the cUTI Arms: 28-34 calendar days from randomization
Population: Extended microbiologically evaluable at FU2
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 0 | 0 | 115 | 117
Participant
  Escherichia coli - Favorable (n=44, 50) |  |  | 28 | 39
  Escherichia coli - Unfavorable (n=44, 50) |  |  | 16 | 11
  Kleb. pneumoniae - Favorable (n= 56, 46) |  |  | 33 | 32
  Kleb. pneumoniae - Unfavorable (n=56, 46) |  |  | 23 | 14
  Pseudo. aeruginosa - Favorable (n=4, 11) |  |  | 2 | 9
  Pseudo. aeruginosa - Unfavorable (n=4, 11) |  |  | 2 | 2

32. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at TOC by CAZ-AVI MIC in mMITT Analysis Set
Description: Proportion of patients with a favorable per-pathogen microbiological response for pathogens (>=10% of frequncy in the combined cIAI and cUTI patients): favourable microbiological response includes: Eradication Absence (or urine quantification less than 10^4 CFU/ml for cUTI patients) of causative pathogen from an appropriately obtained specimen at the site of infection. If the patient was bacteremic at Screening, the bacteremia has also resolved. Presumed eradication where, repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure (specific to cIAI population). For E.coli, MIC available values are: <=0.008, 0.03, 0.06, 0.12, 0.25, 0.5, 1, 2, 8. For K. pneumoniae, MIC available values are: 0.06, 0.12, 0.25, 0.5, 1, 2, 4, 32, >32. For P. aeruginosa, MIC available values are: 2, 4, 8, 16, 32, >32.
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  E. coli (MIC: <=0.008) - Favorable (n=0, 0, 1, 1) | 0 | 0 | 1 | 1
  E. coli (MIC: 0.03) - Favorable (n=0, 0, 0, 2) | 0 | 0 | 0 | 1
  E. coli (MIC: 0.06) - Favorable (n=1, 0, 3, 2) | 0 | 0 | 3 | 2
  E. coli (MIC: 0.12) - Favorable (n=4, 2, 20, 20) | 2 | 1 | 12 | 16
  E. coli (MIC: 0.25) - Favorable (n=0, 0, 15, 16) | 0 | 0 | 10 | 15
  E. coli (MIC: 0.5) - Favorable (n=0, 1, 8, 11) | 0 | 1 | 5 | 10
  E. coli (MIC: 1) - Favorable (n=0, 0, 2, 2) | 0 | 0 | 1 | 2
  E. coli (MIC: 2) - Favorable (n=0, 0, 2, 1) | 0 | 0 | 2 | 1
  E. coli (MIC: 8) - Favorable (n=0, 0, 2, 4) | 0 | 0 | 2 | 4
  K. pneumoniae (MIC: 0.06) - Favorable (n=0,0,2,0) | 0 | 0 | 1 | 0
  K. pneumoniae (MIC: 0.12) - Favorable (n=0,1,8,5) | 0 | 0 | 6 | 4
  K. pneumoniae (MIC: 0.25) - Favorable (n=0,3,12,6) | 0 | 2 | 7 | 5
  K. pneumoniae (MIC: 0.5) - Favorable (n=2,0,24,22) | 1 | 0 | 16 | 19
  K. pneumoniae (MIC: 1) - Favorable (n=0,0,16,18) | 0 | 0 | 11 | 16
  K. pneumoniae (MIC: 2) - Favorable (n=1, 1, 1, 2) | 1 | 1 | 1 | 1
  K. pneumoniae (MIC: 4) - Favorable (n=0, 0, 1, 1) | 0 | 0 | 1 | 0
  K. pneumoniae (MIC: 32) - Favorable (n=0, 0, 1, 0) | 0 | 0 | 0 | 0
  K. pneumoniae (MIC: >32) - Favorable (n=0,0,0,1) | 0 | 0 | 0 | 0
  P. aeruginosa (MIC: 2) - Favorable (n=1, 0, 0, 1) | 1 | 0 | 0 | 1
  P. aeruginosa (MIC: 4) - Favorable (n=0, 0, 3, 2) | 0 | 0 | 1 | 1
  P. aeruginosa (MIC: 8) - Favorable (n=0, 0, 0, 2) | 0 | 0 | 0 | 2
  P. aeruginosa (MIC: 16) - Favorable (n=0, 1, 0, 1) | 0 | 1 | 0 | 0
  P. aeruginosa (MIC: 32) - Favorable (n=0, 0, 1, 3) | 0 | 0 | 1 | 3
  P. aeruginosa (MIC: >32) - Favorable (n=0,0,1,5) | 0 | 0 | 1 | 4

33. Secondary Outcome: Per-pathogen Microbiological Response of Gram-negative Pathogen at TOC by CAZ-AVI MIC in EME at TOC Analysis Set
Description: Proportion of patients with a favorable per-pathogen microbiological response for pathogens (>=10% of frequncy in the combined cIAI and cUTI patients): favourable microbiological response includes: Eradication Absence (or urine quantification less than 10^4 CFU/ml for cUTI patients) of causative pathogen from an appropriately obtained specimen at the site of infection. If the patient was bacteremic at Screening, the bacteremia has also resolved. Presumed eradication where, repeat cultures were not performed/clinically indicated in a patient who had a clinical response of cure (specific to cIAI population). For E.coli, MIC available values are: <=0.008, 0.03, 0.06, 0.12, 0.25, 0.5, 1, 2, 8. For K. pneumoniae, MIC available values are: 0.06, 0.12, 0.25, 0.5, 1, 2, 4, >32. For P. aeruginosa, MIC available values are: 2, 4, 8, 16, 32, >32.
Time Frame: 6-12 days after last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Extended microbiologically evaluable at TOC
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 8 | 124 | 131
Participant
  E. coli (MIC: <=0.008) - Favorable (n=0, 0, 1, 1) | 0 | 0 | 1 | 1
  E. coli (MIC: 0.03) - Favorable (n=0, 0, 0, 2) | 0 | 0 | 0 | 1
  E. coli (MIC: 0.06) - Favorable (n=0, 0, 3, 1) | 0 | 0 | 3 | 1
  E. coli (MIC: 0.12) - Favorable (n=2, 1, 18, 18) | 2 | 1 | 10 | 16
  E. coli (MIC: 0.25) - Favorable (n=0, 0, 13, 15) | 0 | 0 | 9 | 15
  E. coli (MIC: 0.5) - Favorable (n=0, 1, 6, 9) | 0 | 1 | 4 | 9
  E. coli (MIC: 1) - Favorable (n=0, 0, 2, 2) | 0 | 0 | 1 | 2
  E. coli (MIC: 2) - Favorable (n=0, 0, 2, 1) | 0 | 0 | 2 | 1
  E. coli (MIC: 8) - Favorable (n=0, 0, 2, 4) | 0 | 0 | 2 | 4
  K. pneumoniae (MIC: 0.06) - Favorable (n=0,0,1,0) | 0 | 0 | 0 | 0
  K. pneumoniae (MIC: 0.12) - Favorable (n=0,0,8,5) | 0 | 0 | 6 | 4
  K. pneumoniae (MIC: 0.25) - Favorable (n=0,2,11,6) | 0 | 2 | 7 | 5
  K. pneumoniae (MIC: 0.5) - Favorable (n=1,0,23,21) | 1 | 0 | 16 | 19
  K. pneumoniae (MIC: 1) - Favorable (n=0,0,15,17) | 0 | 0 | 11 | 15
  K. pneumoniae (MIC: 2) - Favorable (n=1, 1, 1, 2) | 1 | 1 | 1 | 2
  K. pneumoniae (MIC: 4) - Favorable (n=0, 0, 1, 1) | 0 | 0 | 1 | 0
  K. pneumoniae (MIC: >32) - Favorable (n=0,0,0,1) | 0 | 0 | 0 | 0
  P. aeruginosa (MIC: 2) - Favorable (n=1, 0, 0, 1) | 1 | 0 | 0 | 1
  P. aeruginosa (MIC: 4) - Favorable (n=0, 0, 3, 2) | 0 | 0 | 1 | 1
  P. aeruginosa (MIC: 8) - Favorable (n=0, 0, 0, 2) | 0 | 0 | 0 | 2
  P. aeruginosa (MIC: 16) - Favorable (n=0, 1, 0, 1) | 0 | 1 | 0 | 0
  P. aeruginosa (MIC: 32) - Favorable (n=0, 0, 1, 3) | 0 | 0 | 1 | 3
  P. aeruginosa (MIC: >32) - Favorable (n=0,0,1,4) | 0 | 0 | 1 | 4

34. Secondary Outcome: The Reason for Treatment Change/Discontinuation in mMITT Analysis Set
Description: Proportion of patients in the mMITT analysis set for whom the assigned study treatment was changed, discontinued, or interrupted. Creatinine clearance (CrCl)
Time Frame: From first infusion to last infusion of study therapy. Duration of study therapy was 5 to 21 days.
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  Treatment Change | 1 | 0 | 8 | 11
  Treatment Change - Crcl change | 1 | 0 | 5 | 10
  Treatment Change - Other | 0 | 0 | 3 | 1
  Treatment discontinuation | 4 | 0 | 3 | 1
  Treatment discontinuation - AE | 1 | 0 | 1 | 1
  Treatment discontinuation - Other | 3 | 0 | 2 | 0
  Treatment interrupted | 0 | 0 | 0 | 1
  Treatment interrupted - Change of infusion site | 0 | 0 | 0 | 1

35. Secondary Outcome: The 28 Days All Cause Mortality Rate in mMITT Analysis Set
Description: Proportion of patients with Day 28 all-cause mortality in mMITT analysis set. The death in the cIAI patient were reviewed independently by the SRP Chair.
Time Frame: From first infusion to Day 28
Population: Microbiological modified intent to treat
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 11 | 10 | 137 | 144
Participant
  All cause mortality | 1 | 0 | 3 | 3
  Deaths due to disease progression | 0 | 0 | 0 | 0
  Number of patients with any AE with outcome=death | 1 | 0 | 3 | 3

36. Secondary Outcome: The 28 Days All Cause Mortality Rate in EME at TOC Analysis Set
Description: Proportion of patients with Day 28 all-cause mortality in EME at TOC analysis set. The death in the cIAI patient were reviewed independently by the SRP Chair.
Time Frame: From first infusion to Day 28
Population: Extended microbiologically evaluable at TOC
Measure: Number; unit: Participant
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Number analyzed (Participants) | 5 | 8 | 124 | 131
Participant
  All cause mortality | 0 | 0 | 1 | 1
  Deaths due to disease progression | 0 | 0 | 0 | 0
  Number of patients with any AE withoutcome=death | 0 | 0 | 1 | 1

37. Secondary Outcome: Plasma Concentrations for Ceftazidime and Avibactam - cIAI in PK Analysis Set
Description: Blood samples were taken on Day 3 for ceftazidime and avibactam plasma concentration.
Time Frame: Anytime within 15 minutes prior to or after stopping study drug, anytime between 30 to 90 minutes after stopping study drug, anytime between 300 to 360 minutes after stopping study drug
Population: PK Analysis set
Measure: Geometric Mean (Full Range); unit: NG/ML
Groups:
- CAZ (1); AVI (1): 15 mins before/after dose
- CAZ (2); AVI (2): 30-90 mins after dose
- CAZ (3); AVI (3): 300-360 mins after dose
Arm/Group | CAZ (1) | AVI (1) | CAZ (2) | AVI (2) | CAZ (3) | AVI (3)
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
NG/ML | 23880.3 [2700 to 80900] | 3061.3 [286 to 13200] | 39465.3 [2620 to 85500] | 6304.1 [285 to 15500] | 14904.8 [2500 to 58100] | 1769.3 [277 to 7900]

38. Secondary Outcome: Plasma Concentrations for Ceftazidime and Avibactam - cUTI in PK Analysis Set
Description: Blood samples were taken on Day 3 for ceftazidime and avibactam plasma concentration.
Time Frame: as for outcome 37
Population: PK Analysis set
Measure: Geometric Mean (Full Range); unit: NG/ML
Arm/Group | CAZ (1) | AVI (1) | CAZ (2) | AVI (2) | CAZ (3) | AVI (3)
Number analyzed (Participants) | 145 | 147 | 141 | 147 | 146 | 146
NG/ML | 74260.2 [5970 to 1640000] | 10103.8 [504 to 376000] | 56905.9 [14700 to 1910000] | 8141.2 [773 to 405000] | 21442.0 [2490 to 1600000] | 2425.0 [315 to 431000]

ADVERSE EVENTS:
Time Frame: Non serious AEs and SAEs were from the first infusion of study therapy through the FU visits (cIAI: 28-35 days calendar days from randomization, cUTI: 28-32 calendar days from randomization).
Description: One participant in the "cUTI:CAZ-AVI" arm was randomized but did not receive study drug. This participant was not included in the safety analysis."
Arm/Group | cIAI:Best Available Therapy | cIAI:CAZ-AVI + Metronidazole | cUTI:Best Available Therapy | cUTI:CAZ-AVI
Serious Adverse Events (participants affected / at risk) | 5/15 | 2/12 | 5/153 | 7/152
Other Adverse Events (participants affected / at risk) | 12/15 | 8/12 | 36/153 | 18/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cIAI:Best Available Therapy (N=15) | cIAI:CAZ-AVI + Metronidazole (N=12) | cUTI:Best Available Therapy (N=153) | cUTI:CAZ-AVI (N=152)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cIAI:Best Available Therapy (N=15) | cIAI:CAZ-AVI + Metronidazole (N=12) | cUTI:Best Available Therapy (N=153) | cUTI:CAZ-AVI (N=152)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 0 (0) | 4 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 8 (8) | 3 (4)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 9 (9) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (5)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (8)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endoscopy gastrointestinal abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 11 (17) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to use such Confidential study information and not to disclose them to any other third parties, except that the undersigned shall not be prevented from using or disclosing information: (a) which by written records was previously known; (b) which is now public knowledge, (c) which is lawfully obtained by the undersigned from sources who have a lawful right to disclose such information.